CLINICAL TRIAL: NCT05325203
Title: A Randomized, Double-blind, Placebo-controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of Recombinant Humanized Anti-PCSK9 Monoclonal Antibody Injection in Subjects With Heterozygous Familial Hypercholesterolemia
Brief Title: A Study to Evaluate the Efficacy and Safety of JS002 in Patients With Heterozygous Familial Hypercholesterolemia (HeFH).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JS002-005
Record Dates: First submitted 2022-02-08; First posted 2022-04-13 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2022-02

CONDITIONS: Heterozygous Familial Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- JS002 150mg Q2W for 24 weeks (Experimental): 40 patients will be enrolled in this arm
  Interventions: Biological: Ongericimab
- placebo 150mg Q2W for 24 weeks (Placebo Comparator): 20 patients will be enrolled in this arm
  Interventions: Drug: Placebo
- JS002 450mg Q4W for 24 weeks (Experimental): 40 patients will be enrolled in this arm
  Interventions: Biological: Ongericimab
- placebo 450mg Q4W for 24 weeks (Placebo Comparator): 20 patients will be enrolled in this arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Ongericimab — Administered by subcutaneous injection
  Other Names: JS002
  Arms: JS002 150mg Q2W for 24 weeks; JS002 450mg Q4W for 24 weeks
Drug: Placebo — Administered by subcutaneous injection
  Arms: placebo 150mg Q2W for 24 weeks; placebo 450mg Q4W for 24 weeks

SUMMARY:
JS002 is a recombinant human anti-PCSK9 monoclonal antibody.The study is a multicenter, randomized, double-blind, placebo-controlled Phase III clinical study in Chinese patients with heterozygous familial hypercholesterolemia (HeFH). Objective To evaluate the efficacy and safety of JS002 150 mg (Q2W) and 450 mg (Q4W) subcutaneous injection (SC).

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled Phase III clinical study evaluating the efficacy and safety of JS002 in patients with heterozygous familial hypercholesterolemia. 120 subjects are planned to be enrolled. Each subject is required a maximum of 6 weeks of screening, 24 weeks of treatment, and 8 weeks of follow-up. To evaluate the lipid-lowering efficacy of subcutaneous injection of JS002 at 24 weeks compared with placebo in heterozygous familial hypercholesterolemia patients under optimized lipid lowing therapy . Subjects meeting the study inclusion criteria will be randomly assigned in a 2:1:2:1 ratio to JS002 150 mg Q2W or JS002 450 mg Q4W or matched placebo to receive the study drug (JS002) or placebo subcutaneously for 24 weeks.

treatment cohorts: JS002 150mg Cohort:JS002 150mg or placebo treatment(JS002 :Placebo=2:1) Q2W JS002 450mg Cohort:JS002 450mg or placebo treatment(JS002 :Placebo=2:1)Q4W

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Males and females ≥ 18 to ≤ 80 years of age
3. DLCN>8 in HeFH
4. Stable lipid-lowering therapies for at least 4 weeks
5. Patients with ASCVD LDL cholesterol≥1.4mmol/L at screening Patients without ASCVD LDL cholesterol≥2.6mmol/L at screening
6. Triglyceride≤4.5 mmol/L（400 mg/dL）;

Exclusion Criteria:

1. HoFH or meet the diagnostic criteria of HoFH
2. New York Heart Association (NYHA) class III or IV or last known left ventricular ejection fraction < 30%
3. History of uncontrolled arrhythmia within 90 days
4. Myocardial infarction, unstable angina, percutaneous coronary intervention (PCI), coronary artery bypass graft (CABG) or stroke within 90 days of randomization
5. Planned cardiac surgery or revascularization.
6. Uncontrolled diabetes mellitius (HbA1c>8.0%）.
7. Uncontrolled hypertension.
8. Other conditions that the researchers considered inappropriate to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2021-12-31 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
Percent Change From Baseline in Low-Density Lipoprotein Cholesterol (LDL-C) at Week 24 | Baseline and week 24
  LDL-C was quantified using the enzymatic colorimetric assay

SECONDARY OUTCOMES:
Absolute Change From Baseline in Low-Density Lipoprotein Cholesterol (LDL-C) at Week 24 | Baseline and Week 24
  LDL-C was quantified using the enzymatic colorimetric assay
Percentage changes From Baseline in the Total Cholesterol at week 24 | Baseline and Week 24
  TC was quantified using the enzymatic colorimetric assay
Absolute changes From Baseline in the Total Cholesterol at week 24 | Baseline and Week 24
  TC was quantified using the enzymatic colorimetric assay
Percentage changes From Baseline in Non-HDL-C at Week 24 | Baseline and Week 24
  Non-HDL-C was quantified using the Calculation,TC minus HDL-C
Absolute changes From Baseline in Non-HDL-C at Week 24 | Baseline and Week 24
  Non-HDL-C was quantified using the Calculation,TC minus HDL-C
Percentage changes From Baseline in Apo B at Week 24 | Baseline and Week 24
  Apo B was quantified using the turbidimetric immunoassay(TIA)
Absolute changes From Baseline in Apo B at Week 24 | Baseline and Week 24
  Apo B was quantified using the turbidimetric immunoassay(TIA)
Percentage changes From Baseline in Lp(a) at Week 24 | Baseline and Week 24
  Lp(a) was quantified using the turbidimetric immunoassay(TIA)
Absolute changes From Baseline in Lp(a) at Week 24 | Baseline and Week 24
  Lp(a) was quantified using the turbidimetric immunoassay(TIA)
Percentage changes From Baseline in HDL-C at Week 24 | Baseline and Week 24
  HDL-C was quantified using the enzymatic colorimetric assay
Absolute changes From Baseline in HDL-C at Week 24 | Baseline and Week 24
  HDL-C was quantified using the enzymatic colorimetric assay
Percentage changes From Baseline in Apo A1 at Week 24 | Baseline and Week 24
  Apo A1 was quantified using the turbidimetric immunoassay(TIA)
Absolute changes From Baseline in Apo A1 at Week 24 | Baseline and Week 24
  Apo A1 was quantified using the turbidimetric immunoassay(TIA)
Percentage changes From Baseline in TG at Week 24 | Baseline and Week 24
  TG was quantified using the enzymatic colorimetric assay
Absolute changes From Baseline in TG at Week 24 | Baseline and Week 24
  TG was quantified using the enzymatic colorimetric assay
The ratio of TC/HDL - C | Baseline and Week 24
  Calculation
The ratio of Apo B/Apo A1 | Baseline and Week 24
  Calculation
Percentage of Participants With 50% or Greater Reduction in LDL-C From Baseline at Week 24 | Baseline and Week 24
  Calculation

OTHER OUTCOMES:
Number of subjects who develop detectable anti-drug antibodies (ADAs) | from baseline to 32 weeks
  ADA was quantified using the Bridging-ECLIA

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital Capital Medical University City:Beijing, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Lin J, Ji Y, Wang G, Ma X, Yao Z, Han X, Chen J, Chen J, Huang W, Xu G, Peng D, Yan P, Qiao P, He Y, Tang Y, Wang M, Zhang M, Yu J, Hao Y, Ma C. Efficacy and safety of ongericimab in Chinese patients with heterozygous familial hypercholesterolemia: A randomized, double-blind, placebo-controlled phase 3 trial. Atherosclerosis. 2025 Apr;403:119120. doi: 10.1016/j.atherosclerosis.2025.119120. Epub 2025 Jan 29. PMID 39999660